CLINICAL TRIAL: NCT04811885
Title: The Effects of Covid-19 Pandemic on the Cardiovascular Heath of Children With Autism
Brief Title: The Effects of Covid-19 Pandemic on the Cardiovascular Heath of Children With Autism Spectrum Disorder
Acronym: ASD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institute of Technology, Carlow (Other)
Responsible Party: Principal Investigator, Katie White, Post graduate research student, Institute of Technology, Carlow
Other Study IDs: Institute Technology Carlow
Record Dates: First submitted 2021-03-02; First posted 2021-03-23 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder; Cardiovascular Health
Keywords: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- child with ASD of school going age: Questionnaire complete by parent with children with ASD semi structure interview complete by parent with children
  Interventions: Other: The Effects of Covid 19 Pandemic on the Cardiovascular Heath of Children With Autism Spectrum Disorder

INTERVENTIONS:
Other: The Effects of Covid 19 Pandemic on the Cardiovascular Heath of Children With Autism Spectrum Disorder — The Effects of Covid 19 Pandemic on the Cardiovascular Heath of Children With Autism Spectrum Disorder
  Other Names: Questionnaire study; Interview study

SUMMARY:
The aim of the questionnaire and semi structured interview was to understand how the Covid 19 pandemic has impacted the cardiovascular health, physical activity levels, sedentary behavior, sleep, anxiety levels and eating habits of children with ASD in comparison to before the pandemic.

DETAILED DESCRIPTION:
A questionnaire was designed and was available for completion on the colleges survey monkey account. The link for the questionnaire and an explanation of the purpose of the questionnaire was e-mailed to relevant Autism charities or groups within Ireland, the UK and the USA and the administrators of these group were requested to send the link for the questionnaire onto their members. The administrators of relevant social media sites such as Facebook Autism groups were contacted and asked for permission to share the link for the questionnaire to be circulated on their Facebook page.

The questionnaire was completed by parents of children with ASD and consisted of questions relating to them and their child. Within the questionnaire they were asked about their socio-economic background and about their ASD child's cardiovascular health, physical activity levels, sedentary behavior, eating habits and anxiety levels during the Covid 19 pandemic compared to normal life before the outbreak of the pandemic. The aim of the questionnaire was to understand how the Covid 19 pandemic has impacted the cardiovascular health, physical activity levels, sedentary behavior, sleep, anxiety levels and eating habits in comparison to before the pandemic.

The questionnaires was completed online through IT Carlow's survey monkey. Individual results were anonymous and results of the questionnaire were stored on a password protected computer. Participants completed a consent form that explained that participation in the survey was completely voluntary and they could withdraw at any stage if they wished to do so. If they did not wish to answer a question, was a prefer not to say option available and they could continue with the survey. Parents had an option at the end of the survey to enter their email address which allowed them to partake in any follow up questionnaire studies. The questionnaire was initially piloted and was amended as necessary based on the results of the pilot study.

The second aspect will of the study used qualitative design (semi-structured interviews, n=10) to gain deeper insights into the challenges and barriers to engaging children with autism in healthy lifestyle behaviours and the effects COVID 19 had on these challenges and barriers. Each interview was approximately 60 minutes in length. A semi-structured, qualitative interview schedule, which is attached below guided the interview process and was continually revised based on reflection and evolving conceptualisation. Written consent was sought from all participants. The consent form explained that participation in the interview was completely voluntary and they could withdraw at any stage if they wished to do so. If they did not wish to answer a question, they could decline and move on to the next question. The interview was initially piloted and was amended as necessary based on the results of the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* children with ASD

Exclusion Criteria:

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: child with ASD of school going age living in Ireland, UK and USA.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-10-14 (Estimated); Study Completion 2021-10-14 (Estimated)

PRIMARY OUTCOMES:
The Effects of Covid-9 Pandemic on the Cardiovascular Heath of Children With Autism Spectrum Disorder | 24 months
  Questionnaire, interview

CONTACTS AND LOCATIONS:
Overall Officials: Katie White, Principal Investigator — Institute of Technology, Carlow
Locations (1):
- Institute of Technology Carlow, Carlow, Lenister, Ireland

IPD SHARING:
Plan to Share IPD: Undecided